CLINICAL TRIAL: NCT01973387
Title: A Randomized, Multicenter, Open-Label, Phase 3 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor PCI-32765 (Ibrutinib) Versus Rituximab in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study of PCI-32765 (Ibrutinib) Versus Rituximab in Relapsed or Refractory Chronic Leukemia/Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR102604; PCI-32765CLL3002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic lymphocytic leukemia; Small lymphocytic lymphoma; Relapsed or refractory chronic lymphocytic leukemia; Relapsed or refractory small lymphocytic lymphoma; Ibrutinib; PCI-32765; Bruton's tyrosine kinase inhibitor; Rituximab; Asia Pacific region participants
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Rituximab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Experimental)
  Interventions: Drug: Rituximab
- Treatment Arm B (Experimental)
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Rituximab — Up to 6 cycles (total of 8 doses administered by intravenous infusion): 375 mg/m2 on Day 1 of Cycle 1, 500 mg/m2 on Day 15 of Cycle 1 (Weeks 1-4); 500 mg/m2 on Day 1 and Day 15 of Cycle 2 (Weeks 5-8); and 500 mg/m2 on Day 1 of Cycles 3-6 (Weeks 9-24).
  Arms: Treatment Arm A
Drug: Ibrutinib — 420 mg capsules administered by mouth daily until disease progression or unacceptable toxicity, whichever occurs first.
  Arms: Treatment Arm B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ibrutinib versus rituximab in adult Asia Pacific region patients with relapsed or refractory chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL).

DETAILED DESCRIPTION:
This is a randomized (individuals assigned to study treatment by chance), open-label (identity of assigned study drug will be known) study designed to evaluate the efficacy and safety of ibrutinib versus rituximab in adult Asia Pacific region patients with relapsed/refractory CLL or SLL with active disease requiring treatment who have failed at least 1 prior line of therapy and are not considered appropriate candidates for treatment or retreatment with purine analog-based therapy. Approximately 150 patients will be randomly assigned in a 1:2 ratio into 2 treatment arms to receive either intravenous rituximab (Treatment Arm A) for 6 cycles or oral ibrutinib (Treatment Arm B) until disease progression or unacceptable toxicity, whichever occurs first. The study will include screening, treatment, and follow-up phases. Treatment will extend from randomization until study drug discontinuation. Follow-up will consist of 2 phases: post-treatment (from the discontinuation of treatment for reasons other than disease progression until the patient has progressive disease) and post-disease progression (subsequent anticancer therapy and survival status will be recorded until death, lost to follow-up, consent withdrawal, or study closure). Patients in the rituximab arm with disease progression or who meet the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria for requiring subsequent anti-CLL therapy may be considered for cross over to receive ibrutinib 420 mg orally, daily until disease progression, unacceptable toxicity, withdrawal from study, or until study end whichever occurs earliest. Efficacy evaluations will assess for disease response and progression in accordance with International Workshop on Chronic Lymphocytic Leukemia 2008 criteria. Serial pharmacokinetic (study of what a drug does to the body) blood samples will be collected in the ibrutinib treatment group. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status of 0-1
* Diagnosis of chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL) that meets protocol-defined criteria
* Laboratory values within protocol-defined parameters
* Active disease meeting International Workshop on Chronic Lymphocytic Leukemia 2008 criteria
* Received at least 1 prior therapy for CLL/SLL and not appropriate for treatment or retreatment with purine analog-based therapy
* Measurable nodal disease by computed tomography
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test at Screening and agree to use highly effective methods of contraception during the study and for 90 days following the last dose with ibrutinib or 12 months following the last dose of rituximab

Exclusion Criteria:

* Central nervous system lymphoma or leukemia
* Prolymphocytic leukemia or history of or currently suspected Richter's transformation
* Refractory to prior rituximab-based therapy
* Received any chemotherapy, external beam radiation therapy, anticancer antibodies, or investigational drug within 30 days prior to first dose of study drug
* Corticosteroid use >20 mg within 1 week prior to first dose of study drug
* Radio- or toxin-conjugated antibody therapy within 10 weeks prior to first dose of study drug
* Prior autologous transplant within 6 months prior to first dose of study drug
* Prior allogeneic stem cell transplant
* Major surgery within 4 weeks prior to first dose of study drug
* History of prior malignancy according to protocol-defined criteria
* Currently active clinically significant cardiovascular disease within 6 months prior to first dose with study drug
* Uncontrolled active systemic fungal, bacterial, viral, or other ongoing anti-infective treatment administered intravenously
* History of human immunodeficiency virus or active infection with hepatitis B or C
* History of stroke or intracranial hemorrhage within 6 months prior to random assignment
* Pregnant or lactating women
* Current life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, or put the study at risk
* Requires or receiving anticoagulation with warfarin or equivalent Vitamin K antagonists
* Requires treatment with a strong CYP3A4/5 inhibitor
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP), defined as declining hemoglobin or platelet count secondary to autoimmune destruction within the screening period or requirement for high doses of steroids (greater than [>]20 milligram [mg] daily of prednisone daily or equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2017-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (26):
- Australia (5):
  - Concord
  - Gosford
  - Heidelberg
  - Perth
  - Tweed Heads
- China (13):
  - Beijing
  - Chendu
  - Fuzhou
  - Guangzhou
  - Jinan
  - Nanjing
  - Qingdao
  - Shanghai
  - Suzhou
  - Tianjin
  - Unk Hangzhou
  - Wuhan
  - Xi'an
- Malaysia (4):
  - Johor Bahru
  - Kuala Lumpur
  - Malacca
  - Subang Jaya
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Tainan
  - Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Randomized, Multicenter, Open-Label, Phase 3 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor PCI-32765 (Ibrutinib) versus Rituximab in Subjects with Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Groups:
- Ibrutinib: Receive 420 mg ibrutinib (3 x 140-mg capsules) by mouth once daily continuous (without interruption) self-administered home treatment until disease progression or unacceptable toxicity, whichever occurs first.
- Rituximab: Receive rituximab IV infusion 375 mg/m2 on Day 1 of Cycle 1 and 500 mg/m2 on Day 15 of Cycle 1 (Weeks 1-4); 500 mg/m2 on Day 1 and Day 15 of Cycle 2 (Weeks 5-8); 500 mg/m2 on Day 1 of Cycles 3-6 (Weeks 9-24).
Period: Overall Study
Arm/Group | Ibrutinib | Rituximab
Started | 106 | 54
Treated | 104 | 52
Completed | 0 | 36
Not Completed | 106 | 18
Not completed — Adverse Event | 14 | 4
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Study terminated by sponsor | 63 | 0
Not completed — Progressive disease or relapse | 16 | 5
Not completed — Death | 4 | 3
Not completed — Randomized, not treated | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrutinib | Rituximab | Total
Number analyzed (Participants) | 106 | 54 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (10.36) | 63.6 (13.04) | 63.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 18 | 47
  Male | 77 | 36 | 113
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 15 | 9 | 24
  China | 87 | 44 | 131
  Malaysia | 1 | 1 | 2
  Taiwan, Province Of China | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the interval between the date of randomization and the date of disease progression or death, whichever was first reported. International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria for progressive disease (PD): New enlarged nodes greater than (>)1.5 centimeter (cm), new hepatomegaly or splenomegaly, or other organ infiltrates; greater than or equal to (>=)50 percent (%) increase from nadir in existing lymph node or >=50% increase from nadir in sum of product of diameters of multiple nodes; >=50% increase from nadir in enlargement of liver or spleen; >=50% increase from baseline in lymphocyte count (and to >=5*10^9/L) unless considered treatment-related lymphocytosis; New cytopenia (Hemoglobin b [Hgb] or platelets) attributable to chronic lymphocytic leukemia (CLL) and transformation to a more aggressive histology.
Time Frame: From the date of randomization to the date of disease progression or death, whichever was first reported (Up to 3.7 years)
Population: Intent-to-Treat (ITT) analysis set is defined as all participants randomized into the study and analyzed according to assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ibrutinib: Treatment Arm A received 420 milligram (mg) ibrutinib (3*140-mg capsules) by mouth once daily continuous (without interruption) self-administered home treatment until disease progression or unacceptable toxicity, whichever occurs first.
- Rituximab: Treatment Arm B received rituximab intravenous (IV) infusion 375 milligrams per meter square (mg/m^2) on Day 1 of Cycle 1 and 500 mg/m^2 on Day 15 of Cycle 1 (Weeks 1-4); 500 mg/m^2 on Day 1 and Day 15 of Cycle 2 (Weeks 5-8); 500 mg/m^2 on Day 1 of Cycles 3-6 (Weeks 9-24).
Arm/Group | Ibrutinib | Rituximab
Number analyzed (Participants) | 106 | 54
months | NA [NA to NA] — Median, lower limit and upper limit of 95% CI was not estimable due to lesser number of events. | 8.38 [8.31 to 9.03]
Statistical Analysis 1: Comparison: Ibrutinib vs Rituximab; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.178, 95% CI 2-sided [0.109 to 0.291]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR defined as number of participants achieving a complete response (CR), complete response with incomplete marrow recovery (CRi), nodular partial response (nPR) or partial response (PR). IWCLL 2008 criteria: CR- No lymphadenopathy and hepatosplenomegaly, no constitutional symptoms, neutrophils >1.5*10^9/liter (L), platelets >100*10^9/L, Hgb >11 gram per deciliter (g/dL) and absolute lymphocyte count <4000/microliter (mcL); CRi- CR with incomplete recovery of bone marrow; nPR- participants meet criteria for CR, but the bone marrow biopsy shows B-lymphoid nodules, may represent a clonal infiltrate; PR- >=50% drop in lymphocyte count from baseline or <=4.0*10^9/L with following: >=50% decrease in sum products of up to 6 lymph nodes, no new enlarged lymph nodes, When abnormal, >=50% decrease in enlargement of spleen from baseline or normalization and a response in 1 of following: Neutrophils >1.5*10^9/L, Platelets>100000/mcL and Hgb>11 g/dL or >=50% improvement over baseline in all.
Time Frame: From the date of randomization to disease progression (Up to 3.7 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ibrutinib | Rituximab
Number analyzed (Participants) | 106 | 54
participants | 66 | 4

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the interval between the date of randomization and the date of death from any cause.
Time Frame: From the date of randomization to the date of death (Up to 3.7 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib | Rituximab
Number analyzed (Participants) | 106 | 54
months | NA [NA to NA] — Median, upper limit and lower limit of 95% CI was not estimable due to lesser number of events. | NA [19.52 to NA] — Median and upper limit of 95% CI was not estimable due to lesser number of events.

4. Secondary Outcome: Number of Participants With Sustained Hematologic Improvement
Description: Sustained hematologic improvement was defined as hematological improvement that was sustained continuously for greater than or equal to (>=) 56 days without blood transfusion or growth factors: 1) Platelet counts greater than (>)100* 109/liter (L) if baseline less than or equal to (<=) 100*109/L or increase >= 50 percent (%) over baseline; 2) Hemoglobin >11 gram per deciliters (g/dL) if baseline <= 11 g/dL or increase >= 2 g/dL over baseline.
Time Frame: From the date of randomization to disease progression (Up to 3.7 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ibrutinib | Rituximab
Number analyzed (Participants) | 106 | 54
participants
  Hemoglobin | 43 | 14
  Platelets | 48 | 12

5. Secondary Outcome: Number of Participants With Clinically Relevant Shifts in Disease-Related Symptoms
Description: The most common disease-related symptoms associated with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) (fatigue, weight loss, fevers, night sweats, and abdominal discomfort/splenomegaly) were reported by grade.
Time Frame: From the date of randomization to disease progression (Up to 3.7 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Ibrutinib | Rituximab
Number analyzed (Participants) | 106 | 54
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening up to follow up phase (approximately 3.7 years)
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Ibrutinib | Rituximab
All-Cause Mortality (participants affected / at risk) | 21/104 | 20/52
Serious Adverse Events (participants affected / at risk) | 56/104 | 17/52
Other Adverse Events (participants affected / at risk) | 103/104 | 46/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib (N=104) | Rituximab (N=52)
Agranulocytosis (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 3 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Splenic Infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 3 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 3 | 1
Cardiac Tamponade (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Dry Eye (Eye disorders) | 1 | 0
Eye Irritation (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest Discomfort (General disorders) | 1 | 0
Death (General disorders) | 3 | 0
Local Swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 1
Anal Abscess (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Herpes Virus Infection (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Infected Cyst (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 2
Infective Exacerbation of Bronchiectasis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lung Abscess (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 12 | 6
Pneumonia (Infections and infestations) | 5 | 1
Pneumonia Viral (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Pyelonephritis Chronic (Infections and infestations) | 1 | 0
Salmonella Sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Septic Shock (Infections and infestations) | 1 | 0
Serratia Bacteraemia (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 2 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 2 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Splenic Rupture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 2 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Richter's Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0
Lacunar Infarction (Nervous system disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Renal Cyst (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Circulatory Collapse (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Varicose Vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib (N=104) | Rituximab (N=52)
Anaemia (Blood and lymphatic system disorders) | 20 | 5
Leukocytosis (Blood and lymphatic system disorders) | 13 | 0
Monocytopenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 26 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 3
Vertigo (Ear and labyrinth disorders) | 13 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 1
Constipation (Gastrointestinal disorders) | 18 | 0
Diarrhoea (Gastrointestinal disorders) | 41 | 4
Mouth Ulceration (Gastrointestinal disorders) | 15 | 3
Nausea (Gastrointestinal disorders) | 18 | 1
Vomiting (Gastrointestinal disorders) | 8 | 3
Chills (General disorders) | 1 | 9
Fatigue (General disorders) | 30 | 6
Oedema Peripheral (General disorders) | 10 | 2
Pyrexia (General disorders) | 27 | 14
Lung Infection (Infections and infestations) | 17 | 3
Nasopharyngitis (Infections and infestations) | 19 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 29 | 7
Contusion (Injury, poisoning and procedural complications) | 6 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 3
Alanine Aminotransferase Increased (Investigations) | 7 | 3
Aspartate Aminotransferase Increased (Investigations) | 6 | 3
Blood Creatinine Increased (Investigations) | 6 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 10 | 1
Haemoglobin Decreased (Investigations) | 15 | 6
Lymphocyte Count Increased (Investigations) | 15 | 0
Neutrophil Count Decreased (Investigations) | 36 | 20
Platelet Count Decreased (Investigations) | 33 | 14
Weight Decreased (Investigations) | 8 | 3
White Blood Cell Count Decreased (Investigations) | 9 | 9
Decreased Appetite (Metabolism and nutrition disorders) | 11 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 0
Dizziness (Nervous system disorders) | 6 | 0
Headache (Nervous system disorders) | 11 | 2
Insomnia (Psychiatric disorders) | 7 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 13 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 31 | 3
Skin Haemorrhage (Skin and subcutaneous tissue disorders) | 11 | 0
Hypertension (Vascular disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.